CLINICAL TRIAL: NCT00184158
Title: Cubital Tunnel Treatment, Evaluation of Conservative and Operative Alternatives
Brief Title: Treatment for Cubital Tunnel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 056-02
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: Cubital Tunnel Syndrome
Keywords: Cubital tunnel; treatment; nerve compression
MeSH Terms: conditions — Cubital Tunnel Syndrome; Neuroma | interventions — Decompression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: decompression — Conservative, simple decompression and nerve transfer

SUMMARY:
The researchers want to find out the best treatment for cubital tunnel. The researchers establish the degree of nerve compression and then the patients are randomised to different treatment alternatives, ranging from conservative to operative treatments.

The study is performed at 5 different hospitals in Norway.

ELIGIBILITY:
Inclusion Criteria:

* Patients with cubital tunnel syndrome

Exclusion Criteria:

* Rheumatoid arthritis (RA)
* Osteoarthrosis
* Varus or valgus deformities at elbow

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2005-01 (Actual); Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
pain

SECONDARY OUTCOMES:
electroneurography (ENG
  electroneurography (ENG) before and after the operation and to see if it is consistent with the patient evaluation.
paresthesia
weakness
patient satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: Vilhjalmur Finsen, Prof, Study Director — National Taiwan Normal University
Locations (1):
- St Olavs Hospital, Trondheim, Norway